CLINICAL TRIAL: NCT04205227
Title: A Phase 1/2A Trial of ENB 003 in Combination with Pembrolizumab in Subjects with Advanced Solid Tumors
Brief Title: ENB003 Plus Pembrolizumab Phase 1b/2a in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ENB Therapeutics, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-003-101 (MK3475-951)
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer; Melanoma; Ovary Cancer; Pancreatic Cancer; Solid Tumor
Keywords: solid tumors
MeSH Terms: conditions — Neoplasms; Melanoma; Ovarian Neoplasms; Pancreatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation and Open Label Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- ENB003 150 ug + Pembrolizumab (Experimental): 150 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 300 ug + Pembrolizumab (Experimental): 300 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 500 ug + Pembrolizumab (Experimental): 500 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 750 ug + Pembrolizumab (Experimental): 750 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 1000 ug + Pembrolizumab (Experimental): 1000 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 2000 ug + Pembrolizumab (Experimental): 2000 ug ENB003 will be administered in combination with a fixed dose of pembrolizumab (200mg). In this treatment arm, ENB003 will be administered during each 21 day cycle, as opposed to every other cycle in early arms
  Interventions: Drug: ENB003; Drug: Pembrolizumab
- ENB003 RP2D from dose escalation + Pembrolizumab (Experimental): The recommended phase 2 dose (RP2D) of ENB003 will be selected from the dose escalation portion of the study and administered in combination with a fixed dose of pembrolizumab (200mg)
  Interventions: Drug: ENB003; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ENB003 — ENB003 is selective Endothelin B Receptor Antagonist
Drug: Pembrolizumab — anti-PD1
  Other Names: KEYTRUDA®, MK-3475

SUMMARY:
First-in Human study evaluating the safety, tolerability and efficacy of ENB003 in combination with Pembrolizumab in solid tumors. The study is separated into two parts. Part A is a 3+3 dose escalation to define the recommended RP2D; this part will include metastatic melanoma, platinum resistant ovarian cancer, and pancreatic cancer patients subjects, but other solid tumors will be allowed. Once the RP2D is selected, the study will be expanded into metastatic melanoma, platinum resistant ovarian cancer, and pancreatic cancer subjects. A small number of sarcoma subjects will be included, as exploratory.

DETAILED DESCRIPTION:
Part A: Dose Escalation (with Run-in) A 7-day run-in period of ENB-003 monotherapy, will be administered to all Part A subjects on Days -7, -5 and -3, prior to initiating combination therapy with pembrolizumab at Day 1. ENB-003 will also be administered on Days 1, 3 and 5 in Cycle 1. In subsequent cycles, ENB-003 will be administered on Days 1, 3, 5, 8, 10, and 12 of alternate 21-day treatment cycles, starting with Cycle 3.

Dose escalation will follow a standard 3+3 design, with the following doses being administered during Part A:

* 150 µg ENB-003
* 300 µg ENB-003
* 500 µg ENB-003
* 750 µg ENB-003
* 1000 µg ENB-003 and 2000 µg ENB-003. For 2000 µg doses and above, ENB003 will be administered every 21 day cycle.

Pembrolizumab will be administered as 200 mg on Day 1 of each 21-day cycle in all Part A cohorts.

Part B: Dose Expansion Twelve (12) subjects with malignant melanoma, ovarian cancer, or pancreatic cancer will receive 1 x 21-day treatment cycle of ENB-003 at the recommended phase 2 dose (RP2D) selected in Part A + pembrolizumab. If dose limiting toxicities (DLT) occur in no more than 3 subjects , Part B will be expanded with an additional 27 subjects, plus 6 additional subjects with sarcoma. A review of efficacy will be conducted by a Data Safety Monitoring Board (DSMB) in Part B once 39 RP2D subjects (including 9 malignant melanoma subjects, 16 ovarian cancer subjects and 14 pancreatic cancer subjects) have completed their scheduled 12 week CT/MRI scans. Upon approval by the DSMB, a maximum of 64 further subjects will be treated at the RP2D.

ELIGIBILITY:
Subjects must fulfill all the following inclusion criteria relevant to their tumor type to be eligible for participation in the study:

Inclusion Criteria

Malignant Melanoma

* Histopathologically confirmed diagnosis of advanced, unresectable or metastatic malignant melanoma.
* Subjects may have received no more than 3 previous lines of systemic anti-cancer therapy for advanced disease.
* Subjects must have progressed on treatment with an anti-PD1/Ligand 1 (L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression as defined by meeting all of the following criteria:
* Has at least six weeks of anti PD-1/L1 exposure with an approved anti-PD-1/L1 mAb.
* Has a best objective response (according to RECIST) of PD or SD < 6 months. If RECIST not performed, must be determined to have clinical progression within 6 months of initial treatment with anti-PD1 / PD-L1.

Ovarian Cancer

* Histologically proven diagnosis of high grade serous, high grade endometroid or clear cell ovarian cancer, fallopian tube or primary peritoneal carcinoma.
* Platinum refractory disease, defined as PD during the administration period of first-line platinum-based chemotherapy. Platinum resistant disease defined as PD within 6 months (182 days) after last receipt of first-line platinum-based chemotherapy.
* Subjects may have received up to 3 previous lines of systemic anti-cancer therapy for advanced disease.
* Ovarian cancer patients must be tested for the MSI phenotype. If subjects have high microsatellite instability (MSI-H) or mismatch-repair deficiency (dMMR) phenotype they must have been previously treated with anti-PD1 and demonstrated either PD or disease stabilization, for less than 6 months as best response.

Pancreatic Cancer

* Histologically confirmed (previously obtained biopsied) metastatic or locally advanced unresectable pancreatic adenocarcinoma or pancreatic adenocarcinoma that is recurrent after resection, including with intraductal papillary mucinous neoplasm.
* Subjects must have previously received and progressed on FOLFIRINOX or a gemcitabine-based regimen for their pancreatic cancer.
* Subjects may have received no more than 2 previous lines of therapy for advanced/metastatic disease.
* Pancreatic cancer patients must be tested for the MSI phenotype. If subjects have high microsatellite instability (MSI-H) or mismatch-repair deficiency (dMMR) phenotype they must have been previously treated with anti-PD1 and demonstrated either PD or disease stabilization for less than 6 months as best response.

Basket Study:

* The first 10 subjects for each indication must be ETBR+.
* Subjects must have progressed on at least one standard of care therapy and must not have received more than 3 prior systemic therapies.

SCC of the Head and Neck

* Histologically confirmed metastatic SCC of the head and neck.
* Subjects must have progressed on treatment with an anti-PD1/Ligand 1 (L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression as defined by meeting all of the following criteria:
* Has at least six weeks of anti PD-1/L1 exposure with an approved anti-PD-1/L1 mAb.
* Has a best objective response (according to RECIST) of PD or SD < 6 months
* If RECIST not performed, must be determined to have clinical progression within 6 months of initial treatment with anti-PD1 / PD-L1.

Triple Negative Breast Cancer

* Histologically proven diagnosis of metastatic TNBC
* TNBC subjects must be tested for PD-L1 expression. For CPS >10, Subjects must have progressed on treatment with an anti-PD1/Ligand 1 (L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression as defined by meeting all of the following criteria:

Has at least six weeks of anti PD-1/L1 exposure with an approved anti-PD-1/L1 mAb.

Has a best objective response (according to RECIST) of PD or SD < 6 months. If RECIST not performed, must be determined to have clinical progression within 6 months of initial treatment with anti-PD1 / PD-L1.

All Subjects:

* Be willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Has a life expectancy of >3 months.
* Must have confirmed slides or a tumor block available prior to dosing.
* Fresh biopsies for ETBR and biomarker analysis are preferred for all subjects, especially those that have superficial (cutaneous or subcutaneous e.g. lymph nodes) primary or metastatic lesions. If obtaining a fresh biopsy is not possible, subjects must have archival tumor tissue obtained within 24 months of Screening and that is suitable for performing IHC and biomarker analyses.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential (WOCBP), where a WOCBP is defined as:
* Not surgically sterile i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy, or
* Not post-menopausal, defined as amenorrhea for ≥ 2 years without an alternative medical cause.

Note: Women with amenorrhea for < 2 years and who are not surgically sterile i.e. tubal ligation, bilateral oophorectomy, or complete hysterectomy will only be considered not to be of reproductive potential if they have a documented follicle stimulating hormone (FSH) value in the postmenopausal range.

* A WOCBP who agrees to follow contraceptive guidance from the date of informed consent and for at least 150 days after the last dose of study treatment.
* A male subject must agree to use contraception from the date of informed consent and for at least 120 days after the last dose of study treatment AND must refrain from donating sperm during this period.
* Has measurable disease per RECIST Version 1.1, defined as at least one lesion that can be accurately measured by CT scan or MRI. Minimum measurement must be ≥10 mm as assessed by the Investigator. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Has adequate organ function, as defined in table below. Specimens must be collected within 3 days prior to the start of study treatment.

System Laboratory Value Hematological

* Absolute neutrophil count (ANC) ≥1500/µL or ≥1500/mm3
* Platelets ≥100 000/µL or ≥100 000/mm3 Hemoglobin ≥90.0 g/L or ≥5.6 mmol/L1 Renal
* Creatinine OR
* Measured or calculated2 creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 ×ULN OR ≥60 mL/min for subject with creatinine levels >1.5 × institutional ULN

Hepatic

* Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for subjects with liver metastases)

Coagulation

* International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless subject is receiving anticoagulant therapy provided PT or aPTT is within therapeutic range of intended use of anticoagulants
* ALT (SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) = aspartate aminotransferase (serum glutamic oxaloacetic transaminase);
* GFR = glomerular filtration rate; ULN = upper limit of normal.

  1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
  2. Creatinine clearance (CrCl) will be calculated using the Cockcroft-Gault equation.

Capable of understanding and complying with protocol requirements.

Exclusion Criteria

Subjects will be excluded if they fulfill any of the following exclusion criteria:

Pregnancy Exclusion

* A WOCBP who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required.
* Is breastfeeding or expecting to conceive or father children within the projected duration of the study, from the day date of informed consent through to 150 days after the last dose of study treatment for females, and 120 days after the last dose of study treatment for males.

Prior/Concomitant Therapy

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter, prior to treatment.

Note: Subjects must have recovered from all AEs due to previous therapies to ≤Grade 1 severity or baseline. Subjects with ≤Grade 2 neuropathy may be eligible at Investigator's discretion. Subjects with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the surgery prior to starting study treatment, as determined by the Investigator.

* Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis. Note: Subjects must have recovered from all radiation-related toxicities, and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

Prior/Concurrent Clinical Study Experience

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Subjects who have entered the follow-up phase of an investigational study may participate provided it has been 4 weeks after the last dose of the previous investigational agent.

Diagnostic Assessments

* Average Fridericia-corrected QT interval (QTcF) >460 msec for males and QTcF >480 msec for females as measured by electrocardiogram (ECG) at Screening.
* A family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Subjects with basal cell carcinoma of the skin, SCC of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.

* Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Has severe hypersensitivity (≥ Grade 3) to ENB-003 and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Subjects with known human immunodeficiency virus (HIV), active HBV or active HCV infections. Subjects who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to starting treatment (Note: Subjects should remain on HBV antiviral therapy throughout the study and follow local guidelines for HBV anti-viral therapy post completion of the study intervention).

Subjects with a history of HCV infection are eligible if HCV viral load is undetectable at screening (Note: must have completed curative anti-viral therapy at least 4 weeks prior to starting treatment).

* Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
* History of myocardial infarction ≤ 6 months prior to Screening, or uncontrolled congestive heart failure or uncontrolled atrial fibrillation or uncontrolled ventricular arrythmia.
* Has a history of Pulmonary Arterial Hypertension or Renovascular Hypertension
* Blood pressure ≥ (greater than or equal to)150/90 mm Hg.

Other Exclusions

* Has had an allogenic tissue/solid organ transplant.
* Has previously participated in this protocol [ENB-003-101 (MK3475-951)] i.e. a subject previously enrolled in Part A cannot participate in Part B.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of Treatment-Emergent Adverse Events of ENB003 in combination with pembrolizumab, as assessed by NCI CTCAE Version 5 | assessed on every visit while subjects are in the study up to 2 years
  Based on observed or reported AEs. AEs will be evaluated and classified according to NCI CTCAE Version 5.0
Part B: Efficacy of ENB003 in combination with pembrolizumab | up to 2 years while subjects remain in the study
  Melanoma and Ovarian Cancer:
  • ORR, based on RECIST (evaluated in the context of ETBR expression)
Part B: Efficacy of ENB003 in combination with pembrolizumab | up to 2 years while subjects remain in the study
  Pancreatic Cancer:
  • 6-months OS (evaluated in the context of ETBR expression) Note, these outcomes will be measured by tumor type and not in an aggregate as both the futility and final analysis are independently powered for each tumor type

SECONDARY OUTCOMES:
Part B Efficacy Progression-free survival (PFS), | up to 2 years
  defined as time from first dosing to date of first observed progression, based on RECIST, or death from any cause (whichever comes first).
Part B Efficacy: Duration of response | up to 2 years
  based on RECIST
Part B Efficacy: Time to progression | up to 2 years
  defined as time from first dosing to date of first observed progression, based on RECIST
Part B Efficacy: Overall survival | up to 2 years
  defined as time from first dosing to date of death
pharmacokinetic (PK) of ENB-003-AUC | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  AUC, measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
pharmacokinetic (PK) of ENB-003-Cmax | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  Cmax, measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
pharmacokinetic (PK) of ENB-003-Tmax | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  Tmax, measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
pharmacokinetic (PK) of ENB-003-T1/2 | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  t1/2, measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
pharmacokinetic (PK) of ENB-003-Vss | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  Vss measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
pharmacokinetic (PK) of ENB-003-CL | at 05,10,15, 20, 30 45, 60 and 90 minutes, 2 hours, 3 hours, 5 hours, and 8 hours after administration of the ENB003, on Days -7 and -5 during dose escalation and days 1 and 5 during dose expansion
  CL measured through blood samples from 0 up to 8 hrs, for all subjects in the dose escalation and the first 12 subjects in the dose expansion
Exploratory: IHC assessment of ETBR | single sample taken between day 5-8
  changes in immunohistochemistry (IHC) for Endothelin B Receptor (ETBR) based on tissue staining measured as a percent of the tissue sample stained, after administration of ENB-003 in combination with pembrolizumab (for subjects with accessible tumors, in whom biopsies can be safely performed).
Exploratory: IHC assessment of PD-L1 | single sample taken between day 5-8
  changes in immunohistochemistry (IHC) for PDL-1 receptor based on tissue staining measured as a percent of the tissue sample stained, after administration of ENB-003 in combination with pembrolizumab (for subjects with accessible tumors, in whom biopsies can be safely performed).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Cedars Sinai-The Angeles Clinic, Los Angeles, California
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Border Medical Oncology, Albury, New South Wales
  - Blacktown Oncology, Blacktown, New South Wales
  - Kinghorn-St Vincent's Hospital, Darlinghurst, New South Wales

IPD SHARING:
Plan to Share IPD: No